CLINICAL TRIAL: NCT00857532
Title: A Phase 2 Trial of Florbetapir F18 PET Imaging of β-amyloid in Parkinson's Disease Patients With Cognitive Impairment
Brief Title: Florbetapir F 18 PET Imaging of Beta-amyloid in Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A12; 5R43NS063607-02 (NIH)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-02

CONDITIONS: Parkinson's Disease
Keywords: amyloid burden; Parkinson's disease; florbetapir PET; amyloid PET imaging
MeSH Terms: conditions — Parkinson Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal cognitive performance (Experimental): Subjects with age-and education-adjusted standardized Mattis Dementia Rating Scale scores of ≥9, indicating normal cognitive performance.
  Interventions: Drug: florbetapir F 18
- Mild cognitive deficits (Experimental): Subjects with age-and education-adjusted standardized Mattis Dementia Rating Scale scores between 6 and 8, inclusive, indicating mild cognitive deficits.
  Interventions: Drug: florbetapir F 18
- Severe cognitive impairment (Experimental): Subjects with age-and education-adjusted standardized Mattis Dementia Rating Scale scores below 5, indicating moderate to severe cognitive impairment.
  Interventions: Drug: florbetapir F 18

INTERVENTIONS:
Drug: florbetapir F 18 — 10 millicurie (mCi) (370 MBq) florbetapir F 18 Injection
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
The primary aim of this study is to compare regional amyloid burden in Parkinson's disease (PD) to normal control subjects. We hypothesize that there will be significant differences in overall amyloid burden in PD patients compared to age-matched normal controls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be enrolled if they (inclusion criteria):

  * Are males or females ≥60 years of age
  * Meet research diagnostic criteria for Parkinson's disease:
  * Diagnosis of a parkinsonian syndrome

    * Bradykinesia (slowness of initiation of voluntary movement with progressive reduction in speed and amplitude of repetitive actions)
    * At least one of the following: muscle rigidity, rest tremor, postural instability not due to visual, vestibular, cerebellar or proprioceptive causes
  * Supportive criteria for diagnosis of PD (two or more required)

    * Unilateral onset of symptoms and persistent asymmetry
    * Rest tremor present
    * Progressive illness
    * Excellent response to levodopa with dyskinesias
    * Levodopa response for 5 years or more
    * Clinical course of 10 years or more
  * Have the ability to lie flat and tolerate a 10 minute PET scan.

Exclusion Criteria:

* Subjects may not be enrolled if any of the following are present (exclusion criteria):

  * History of repeated strokes, repeated head injury, definite encephalitis
  * Use of neuroleptics at onset of symptoms
  * Sustained remission
  * Strictly unilateral feature persisting > three years after onset
  * Significant supranuclear gaze palsy
  * Cerebellar, pyramidal and early severe autonomic findings
  * Early severe dementia suggesting a diagnosis of dementia with Lewy bodies (DLB)
  * Imaging study showing structural abnormality that could explain parkinsonism
  * Negative response to an adequate levodopa trial
  * Current clinically significant psychiatric disease that prohibits providing informed consent or participation in the study
  * Current clinically significant endocrine or metabolic disease, pulmonary,
  * Women of childbearing potential who are not two or more years post menopausal or surgically sterilized
  * Have received any investigational medications, or have participated in a trial with investigational medications within the last 30 days

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Parkinson's Disease: Subjects with diagnosed Parkinson's Disease received a 370 megabecquerel (MBq) injection of florbetapir F 18 followed by a 10 minute PET scan 50 minutes post-injection.
Period: Overall Study
Arm/Group | Subjects With Parkinson's Disease
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects With Parkinson's Disease: Subjects with diagnosed Parkinson's Disease received a 370 MBq injection of florbetapir F 18 followed by a 10 minute PET scan 50 minutes post-injection.
Arm/Group | Subjects With Parkinson's Disease
Number analyzed (Participants) | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 71.3 (6.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Mean Cortical Amyloid Burden
Description: Standardized uptake value ratios (SUVR) were calculated and compared between subjects with PD and controls. Subjects with Parkinson's Disease (PD) were stratified into one of three groups based on performance on the age and education adjusted Mattis Dementia Rating Scale (DRS-2). The age and education adjusted DRS-2 ranges from 0 (lowest cognitive function) to 20 (highest cognitive function). SUVR is the ratio of tracer uptake in predefined cortical regions, relative to uptake in the whole cerebellum. SUVR values higher than 1 indicate greater amyloid burden in the predefined cortical regions as compared to cerebellum whereas scores less than 1 indicate the opposite. This outcome measure only reports data from the subjects analyzed in this study, the data from normal controls was obtained from a pre-existing database and is not reported here.
Time Frame: 50-60 min after injection
Population: All subjects who were enrolled in the study and received florbetapir scans.
Measure: Mean (Standard Deviation); unit: SUVR
Groups:
- Subjects With Normal Cognitive Performance: Subjects have an age-and education-adjusted standardized Mattis DRS-2 score greater than or equal to 9.
- Subjects With Mild Cognitive Deficits: Subjects have an age-and education-adjusted standardized Mattis DRS-2 score between 6 and 8 inclusive.
- Subjects With Moderate to Severe Cognitive Impairment: Subjects have an age-and education-adjusted standardized Mattis DRS-2 score 5 and below.
Arm/Group | Subjects With Normal Cognitive Performance | Subjects With Mild Cognitive Deficits | Subjects With Moderate to Severe Cognitive Impairment
Number analyzed (Participants) | 12 | 9 | 10
SUVR | 0.990 (0.141) | 1.051 (0.194) | 1.146 (0.237)

2. Secondary Outcome: Correlation Between Global Amyloid Burden and Clinical Measures of Cognitive Decline.
Description: Correlation between amyloid burden (global florbetapir SUVR) and cognitive decline (DRS-2 score) was determined using Spearman's rank order correlation method where SUVR was the dependent variable and the DRS-2 score was the independent variable. This analysis was performed for total DRS-2 score and the five DRS-2 subscale scores. The subscales (score range) are: Attention (0-37), Initiation/Perseveration (0-37), Construction (0-6), Conceptualization (0-39) and Memory (0-25). The total DRS-2 score is the sum of the subscale scores and ranges from 0-144. Higher DRS-2 scores indicate greater cognitive function.
Time Frame: 50-60 min after injection
Population: All subjects who were enrolled in the study and received florbetapir scans.
Measure: Number; unit: Correlation Coefficient
Groups:
- Subjects With Parkinson's Disease: Subjects with diagnosed Parkinson's Disease received a 370 MBq injection of florbetapir followed by a 10 minute PET scan 50 minutes post-injections
Arm/Group | Subjects With Parkinson's Disease
Number analyzed (Participants) | 31
Correlation Coefficient
  Attention | -0.413
  Initiation/Perseveration | -0.332
  Construction | -0.169
  Conceptualization | -0.206
  Memory | -0.263
  DRS-2 Total Score | -0.369
Statistical Analysis 1: Comparison: Subjects With Parkinson's Disease; P-value for "Attention" correlation coefficient. Null hypothesis is that there is no correlation between florbetapir SUVR and DRS-2 attention score; Test type: Superiority or Other; p = 0.021, Spearman's Rank Order Correlation
Statistical Analysis 2: Comparison: Subjects With Parkinson's Disease; P-value for "Initiation/Perseveration" correlation coefficient. Null hypothesis is that there is no correlation between florbetapir SUVR and DRS-2 initiation/perseveration score; Test type: Superiority or Other; p = 0.077, Spearman's Rank Order Correlation
Statistical Analysis 3: Comparison: Subjects With Parkinson's Disease; P-value for "Construction" correlation coefficient. Null hypothesis is that there is no correlation between florbetapir SUVR and DRS-2 construction score; Test type: Superiority or Other; p = 0.364, Spearman's Rank Order Correlation
Statistical Analysis 4: Comparison: Subjects With Parkinson's Disease; P-value for "Conceptualization" correlation coefficient. Null hypothesis is that there is no correlation between florbetapir SUVR and DRS-2 conceptualization score; Test type: Superiority or Other; p = 0.266, Spearman's Rank Order Correlation
Statistical Analysis 5: Comparison: Subjects With Parkinson's Disease; P-value for "Memory" correlation coefficient. Null hypothesis is that there is no correlation between florbetapir SUVR and DRS-2 memory score; Test type: Superiority or Other; p = 0.152, Spearman's Rank Order Correlation
Statistical Analysis 6: Comparison: Subjects With Parkinson's Disease; P-value for "DRS-2 Total" correlation coefficient. Null hypothesis is that there is no correlation between florbetapir SUVR and DRS-2 total score; Test type: Superiority or Other; p = 0.041, Spearman's Rank Order Correlation

3. Secondary Outcome: Correlation of Florbetapir SUVR With CSF Biomarker Values
Description: Correlation between amyloid burden (florbetapir SUVR) and cerebrospinal fluid (CSF) biomarker values (amyloid beta, tau and phospho-tau) was determined using Spearman's rank order correlation in a subset of subjects undergoing CSF analysis where SUVR was the dependent variable and CSF biomarker values were the independent variables.
Time Frame: 50-60 min after injection
Population: Participants were a subset of all subjects enrolled in this study who were also part of an ongoing study looking at the usefulness of CSF biomarkers.
Measure: Number; unit: Correlation Coefficient
Arm/Group | Subjects With Parkinson's Disease
Number analyzed (Participants) | 22
Correlation Coefficient
  Amyloid beta | -0.4387
  Tau | -0.1248
  Phospho-tau | -0.0525
Statistical Analysis 1: Comparison: Subjects With Parkinson's Disease; P-value for "Amyloid beta" correlation coefficient. Null hypothesis is that there is no correlation between florbetapir SUVR and amyloid beta; Test type: Superiority or Other; p = 0.0411, Spearman's Rank Order Correlation
Statistical Analysis 2: Comparison: Subjects With Parkinson's Disease; P-value for "Tau" correlation coefficient. Null hypothesis is that there is no correlation between florbetapir SUVR and tau; Test type: Superiority or Other; p = 0.5800, Spearman's Rank Order Correlation
Statistical Analysis 3: Comparison: Subjects With Parkinson's Disease; P-value for "Phospho-Tau" correlation coefficient. Null hypothesis is that there is no correlation between florbetapir SUVR and phospho-tau; Test type: Superiority or Other; p = 0.8164, Spearman's Rank Order Correlation

ADVERSE EVENTS:
Arm/Group | Subjects With Parkinson's Disease
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 4/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Parkinson's Disease (N=31)
Hypertension (Vascular disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less